CLINICAL TRIAL: NCT02722486
Title: Use of a Vibrotactile Balance Belt System for Vestibular Rehabilitation in the Pediatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jacob Brodsky, Associate in Otolaryngology, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00019992
Record Dates: First submitted 2016-03-04; First posted 2016-03-30 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Vestibular Diseases
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Vestibular Rehabilitation (Active Comparator): Subjects will undergo weekly vestibular rehabilitation sessions for 3 months (a total of 12 sessions of an hour each). During these sessions, standard balance training exercises will be done at the discretion of the physical therapists.
  Interventions: Other: Standard Vestibular Rehabilitation
- Vestibular Rehabilitation/Balance Belt (Experimental): Subjects will undergo weekly vestibular rehabilitation sessions for 3 months (a total of 12 sessions). They will undergo standard balance training exercises with the physical therapists like the control group, but will also undergo an additional 15 minutes of Balance Belt exercises during each session.
  Interventions: Device: Vestibular Rehabilitation/Balance Belt

INTERVENTIONS:
Device: Vestibular Rehabilitation/Balance Belt — With this device, a subject stands on a force platform on the ground, which measures his/her center of pressure. Additionally, there is laptop displaying the video-based exercise programs and a camera that senses the subject's linear sway, roll, and pitch. Information about the subject's position is transmitted via Bluetooth technology to a non-invasive vibrotactile belt which fits comfortably around the subject's waist, over his/her clothing. Using the Sensory Kinetics software, the subject will play a series of games projected on the laptop screen, which prompt him/her to sway in various directions while keeping both feet planted on the force platform.
  Other Names: Sensory Kinetics Balance Rehabilitation System
  Arms: Vestibular Rehabilitation/Balance Belt
Other: Standard Vestibular Rehabilitation — This is the standard three-month vestibular rehabilitation therapy that patients are routinely referred to at Boston Children's Hospital.
  Arms: Standard Vestibular Rehabilitation

SUMMARY:
The investigators aim to compare rehabilitation progress between control patients who will undergo routine vestibular rehabilitation exercises and experimental patients who will undergo exercises using a vibrotactile balance belt (SKBRS - Sensory Kinetics Balance Rehabilitation System) in addition to their routine vestibular rehabilitation regimen during recovery from diseases affecting the vestibular system. The results of this pilot study will help to determine if the vibrotactile balance belt is a useful supplement to traditional vestibular rehabilitation techniques in children suffering from vestibular impairment.

DETAILED DESCRIPTION:
The investigators will conduct a randomized pilot trial to examine the efficacy of the vibrotactile balance belt on vestibular rehabilitation in the pediatric population. All consented patients will be randomly allocated by a statistician to either the experimental group where participants will undergo SKBRS exercises in addition to their routine vestibular rehabilitation regimen, or to the control group where participants will undergo routine vestibular rehabilitation exercises without the SKBRS.

All subjects will undergo weekly vestibular rehabilitation sessions for 3 months (a total of 12 sessions). During these sessions, standard balance training exercises will be done at the discretion of the therapists. Experimental subjects will also undergo 15 minutes of SKBRS exercises during each standard vestibular rehabilitation session. This device uses video-based exercises and a non-invasive vibrotactile belt to measure the subject's position in space and trunk tilt/sway while performing various balance tasks.

All subjects will undergo the following 3 routine tests throughout the course of the therapy to determine their progress: The Balance Error Scoring System (BESS) to measure the subject's static balance, the Clinical Test of Sensory Integration and Balance (CTSIB), an office-based version of the computerized dynamic posturography test, and the Dynamic Gait Index (DGI), which measures dynamic balance. Finally, the investigators will ask all subjects to provide their subjective opinion of their vestibular rehabilitation program and their opinion of the SKBRS by filling out questionnaires.

The primary outcome measure is a comparison of relative balance improvement between subjects who underwent standard vestibular rehabilitation exercises and those who underwent additional therapy with the SKBRS during their rehab sessions. This progress will be measured by the degree of change in the BESS, CTSIB, and DGI scores between subjects' first and final vestibular rehabilitation sessions. The secondary outcome will be the subjects' subjective assessments of the effectiveness of their vestibular rehabilitation (measured by the VRBQ) as well as the experimental subjects' feedback on the SKBRS device (measured by the SKBRS feedback survey).

ELIGIBILITY:
Inclusion Criteria:

* Referred for vestibular rehabilitation due to balance impairment at Boston Children's Hospital.
* English speaking
* Understanding of how to use the device
* Intention to complete full 3 months of vestibular rehabilitation

Exclusion Criteria:

* Patients with developmental delay to a degree that prevents them from understanding how to use the device or that prevents them from being able to provide feedback on their experience with the device.
* Patients who are unable to stand for the 15 minutes necessary to complete the SKBRS exercises

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Change in BESS Score from baseline to 3 months | 0-3 months
  The investigators will measure the change in BESS score between the first vestibular rehabilitation session and the last session (3 months later).
Change in CTSIB Score from baseline to 3 months | 0-3 months
  The investigators will measure the change in CTSIB score between the first vestibular rehabilitation session and the last session (3 months later).
Change in DGI Score from baseline to 3 months | 0-3 months
  The investigators will measure the change in DGI score between the first vestibular rehabilitation session and the last session (3 months later).

SECONDARY OUTCOMES:
Change in subjective symptoms from baseline to 3 months | 0-3 months
  Subjects will fill out validated Vestibular Rehabilitation Benefit Questionnaire before and after 3 months of treatment to determine the change in their subjective dizziness/imbalance symptoms. This will allow the investigators to evaluate the subjective effectiveness of vestibular rehabilitation.
Sensory Kinetics Balance Rehabilitation System Feedback | 3 months
  Experimental subjects will use this questionnaire to give feedback on their experience using the SKBRS. This will be administered on their last visit (3 month point).

CONTACTS AND LOCATIONS:
Overall Officials: Jacob R Brodsky, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital Waltham, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wall C 3rd. Application of vibrotactile feedback of body motion to improve rehabilitation in individuals with imbalance. J Neurol Phys Ther. 2010 Jun;34(2):98-104. doi: 10.1097/NPT.0b013e3181dde6f0. PMID 20588096
- [Background] Wall C 3rd, Wrisley DM, Statler KD. Vibrotactile tilt feedback improves dynamic gait index: a fall risk indicator in older adults. Gait Posture. 2009 Jul;30(1):16-21. doi: 10.1016/j.gaitpost.2009.02.019. Epub 2009 Apr 2. PMID 19345107
- [Background] Wall C 3rd, Oddsson LE, Horak FB, Wrisley DW, Dozza M. Applications of vibrotactile display of body tilt for rehabilitation. Conf Proc IEEE Eng Med Biol Soc. 2004;2004:4763-5. doi: 10.1109/IEMBS.2004.1404318. PMID 17271374
- [Background] Wall C 3rd, Lyford ND, Sienko KH, Balkwill MD. The design and development of a production prototype balance belt. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:3524-8. doi: 10.1109/IEMBS.2011.6090585. PMID 22255100